CLINICAL TRIAL: NCT02106507
Title: Phase 1b Study of ARN 509 Plus Everolimus in Men With Progressive Metastatic Castration-Resistant Prostate Cancer After Treatment With Abiraterone Acetate
Brief Title: ARN 509 Plus Everolimus in Men With Progressive Metastatic Castration-Resistant Prostate Cancer After Treatment With Abiraterone Acetate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Aragon Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-025
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: Apalutamide; RAD001; Everolimus; Castration-resistant; 13-025; ARN-509
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide; Everolimus

ARMS (1):
- Progressive Metastatic Castration-Resistant Prostate Cancer (Experimental): This is a single-institution Phase 1b dose-escalation study in which eligible patients with progressive mCRPC will receive oral doses of apalutamide in combination with everolimus.
  Interventions: Drug: apalutamide; Drug: Everolimus

INTERVENTIONS:
Drug: apalutamide — apalutamide, 240 mg/day, oral
Drug: Everolimus — 5 mg/day of everolimus dose of everolimus will be escalated to 10 mg/day depending on the safety seen during dose escalation and steady-state trough drug levels as recommended

SUMMARY:
The purpose of this study is to test the safety of the combination of apalutamide plus everolimus at different dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate without neuroendocrine differentiation or small cell features with progressive metastatic disease based on any of the following:

  * Rise in PSA: minimum of 3 rising levels, with an interval of at least 1 week between each determination. The last determination must have a value ≥ 2 ng/mL, obtained within 4 weeks of starting study drug, or
  * Measurable disease: new or progressive soft tissue disease on CT or MRI scans, or
  * Radionuclide bone scan: at least 2 new bone lesions, as defined by the PCWG2 criteria1
* Castration-resistant prostate cancer: patients must have surgical or ongoing chemical (androgen deprivation therapy) castration, with baseline testosterone level ≤ 50 ng/dL determined within 4 weeks of starting study drug.
* Dose-Escalation: Prior treatment with abiraterone acetate. At least 4 weeks must have elapsed from the last dose of abiraterone acetate.
* Expansion Cohort only (if conducted in the study): Men with mCRPC and disease progression as defined by PCWG2 within 3 months (primary resistance); or after at least 6 months of treatment (acquired resistance) of starting treatment with abiraterone acetate. At least 4 weeks must have elapsed from the last dose of abiraterone .acetate
* Physiologic doses of corticosteroids are allowed (i.e. no more than 10 mg prednisone daily).
* Patients currently receiving bone loss prevention treatment (e.g. bisphosphonates, denosumab, etc.) must be on a stable dose for at least 4 weeks prior to starting study treatment.
* Patients who received a first generation anti-androgen (e.g., bicalutamide, flutamide, nilutamide) as part of their first-line hormonal therapy must have shown progression of disease off the anti-androgen prior to enrollment.
* At least 4 weeks must have elapsed from the use of androgen receptor antagonists (e.g., bicalutamide, flutamide, nilutamide); 5-α reductase inhibitors (e.g., dutasteride, finasteride, aminoglutethimide); estrogens; ketoconazole and other anti-cancer pharmacologic therapy prior to enrollment.
* At least 6 weeks must have elapsed from the use of bicalutamide if used as part of an initial combined androgen blockage therapy for more than 6 months or if used as second line hormonal therapy and associated with a PSA response of at least 3 months duration.
* At least 12 weeks must have elapsed from the use of Strontium-89, Radium-223 or any investigational or approved immunotherapy (e.g., Provenge) prior to starting study drug.
* At least 4 weeks must have elapsed from the use of any other investigational agent prior to starting study drug.
* At least 4 weeks must have elapsed from major surgery prior to starting study drug.
* Patients with treated, non-progressive epidural disease are eligible.
* At least 18 years of age, with a life expectancy of at least 3 months.
* ECOG performance status 0 or 1 (2 is allowed only if due to bone pain).
* Toxicities related to prior therapy must either have returned to ≤ Grade 1, baseline, or deemed irreversible.
* Physical and laboratory test findings:

  * Adequate hepatic function with serum bilirubin ≤ 1.5 times the upper institutional limits of normal (ULN), ALT and AST ≤ 2.5 x ULN. Patients with a history of Gilbert's syndrome may be enrolled if the total bilirubin is < 3 mg/dL with a predominance of indirect bilirubin
  * Adequate renal function with serum creatinine ≤ 1.5 x ULN
  * Adequate hematologic function with absolute neutrophil counts ≥ 1,500 cells/mm3, platelets ≥ 100,000 cells/mm3 and hemoglobin value ≥ 9 g/dL (Note: patients whose anemia has been corrected to a hemoglobin value ≥ 9 g/dL with blood transfusions are allowed)
  * Electrolytes (including potassium, sodium, and serum calcium corrected for albumin or ionized calcium) must be within normal limits
  * Adequate blood clotting time with an INR <2
* Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* Prior treatment with apalutamide, or PI3K/mTOR pathway inhibitors.
* History of, or current metastases in the brain, meninges, or untreated spinal cord compression.
* Patients previously treated with chemotherapy for mCRPC. At least 12 months must have elapsed from chemotherapy given in the adjuvant or neoadjuvant setting.
* History of any other malignancy within the previous 5 years except for the following: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, stage I or II cancer currently in complete remission, or any other cancer that has been in complete remission for at least 5 years.
* History of seizure or condition that may predispose to seizure (e.g., prior stroke within 1 year of starting study drug, brain arteriovenous malformation)
* Concurrent therapy with medications known to have seizure potential
* Known intolerance or hypersensitivity to Vitamin E, everolimus or to rapamycin derivatives.
* Use of herbal products that may decrease PSA levels (e.g., saw palmetto).
* Known human immunodeficiency virus (HIV) infection.
* Patients who have received live attenuated vaccines within 1 week of start of Everolimus and during the study. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study.
* Patients who are currently part of or have participated in any clinical investigation with an investigational drug within 1 month prior to dosing.
* Male patients whose sexual partner(s) are women of child-bearing potential (WOCBP) who are not willing to use adequate contraception, during the study and for 8 weeks after the end of treatment. Highly effective contraception methods include combination of any two of the following (a+b or a+c or b+c):

  1. Use of oral, injected or implanted hormonal methods of contraception or;
  2. Placement of an intrauterine device (IUD) or intrauterine system (IUS);
  3. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository;
  4. Total abstinence or;
  5. Male/female sterilization.
* Patients with a known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral Everolimus.
* Patients with uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary.
* Patients who have any severe and/or uncontrolled medical conditions such as:

  i. unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤6 months prior to start of Everolimus, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease ii. Symptomatic congestive heart failure of New York heart Association Class III or IV iii. active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable HBV-DNA and/or positive HbsAg, quantifiable HCV-RNA), iv. known severely impaired lung function (spirometry and DLCO 50% or less of normal and O2 saturation 88% or less at rest on room air), v. active, bleeding diathesis;

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
safety | 2 years
  Safety will be evaluated according to the NCI Common Terminology Criteria for Adverse Events V4.0 (CTCAE). Safety assessments will be based on medical review of adverse event reports and the results of vital sign measurements, physical examinations, and clinical laboratory tests throughout the conduct of the study.
pharmacokinetics | 2 years
  Pharmacokinetic parameters (Cmax, Tmax, AUC(INF), AUC(TAU), will be derived from blood to obtain everolimus concentration or plasma to obtain apalutamide and it's major metabolite concentration versus time data for patients in the dose escalation cohorts.
maximum tolerated dose (MTD) | 2 years
  The first phase of the study will examine the safety of apalutamide in combination with everolimus in patients with metastatic castration-resistant prostate cancer. Up to 2 dose levels will be tested. A standard "3 plus 3" dose escalation rule will be used in order to determine the MTD/RP2D. Patients will be treated in cohorts of three and the dosage will be escalated if the clinical toxicity is acceptable. The MTD is defined as the highest dose with an observed incidence of dose limiting toxicity (DLT) in no more than one out of six patients treated at a particular dose level.

SECONDARY OUTCOMES:
anti-tumor activity | 2 years
  Tumor biopsies pre- and post-treatment will be collected to evaluate for downstream indicators of PI3K pathway modulation, including pS6K, p4EBP1, pAKT, AR, PHLLP 1 and 2, and additional pathways of interest if safe and feasible per treating investigator. In lieu of biopsy, if a patient is having an elective or clinical resection/surgery and tissue is already being removed, some of that tissue may be collected for research purposes to fulfill the biopsy requirement for that timepoint. These biomarkers will be measured at baseline and cycle 2 and after treatment to explore the association between changes in the tumor biomarkers and progression-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Rathkopf, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/